CLINICAL TRIAL: NCT05168059
Title: Clevidipine for Acute High Blood Pressure Control in Neurocritical Patients
Brief Title: Clevidipine in Neurocritical Patients
Acronym: NEURO-CLEV
Status: Completed | Type: Observational
Sponsor: Hospital de Cruces (Other)
Collaborators: Biobizkaia Health Research Institute (Other Government)
Responsible Party: Principal Investigator, Blanca Escontrela, Consultant Anesthesiology and Reanimation, Hospital de Cruces
Other Study IDs: CEIC E19/17
Record Dates: First submitted 2021-11-18; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: High Blood Pressure
Keywords: clevidipine; neurocritical
MeSH Terms: conditions — Hypertension | interventions — clevidipine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Clevidipine 0.5 MG/ML Intravenous Emulsion — Effectiveness and safety of clevidipine
  Other Names: CLEVIPREX

SUMMARY:
Acute blood pressure elevation is a frequent problem in neurocritical patients. Its effective management is challenging and must avoid significant decreases of blood pressure leading to lower cerebral perfusion pressure worsening ischemia and elevations probably associated with bleeding, rebleeding or hematoma expansion associated with poor prognosis

DETAILED DESCRIPTION:
Retrospective, observational and single-group study for observe effectiveness and safety of clevidipine for perioperative control of hypertension in patients admitted to Post-Operative Intensive Care Unit after thrombectomy for stroke, intracerebral hemorrhage requiring surgical treatment, embolization of aneurysm after subarachnoid hemorrhage, scheduled neurosurgical and neuroradiology procedures.

ELIGIBILITY:
Inclusion criteria:

1. -Adult patients older than 18 years old admitted to Post-Operative Intensive Care Unit with neurocritical condition requiring surgical or interventional treatment.
2. -Acute High Blood Pressure requiring urgent treatment (SBP ≥160 mmHg or ≥ 20% increase in preoperative values that persists for more than 15 minutes)
3. -Clevidipine used as a first line or after failure of different antihypertensive drugs.

Exclusion criteria:

1. -Adults older than 90 years admitted to Post-Operative Intensive Care Unit with neurocritical condition requiring surgical or interventional treatment.
2. -Patients admitted to Post-Operative Intensive Care Unit with neurocritical condition not requiring surgical or interventional treatment.

Age Groups: Child, Adult, Older Adult
Study Population: Neurocritical patients admitted to PostOperative Intensive Care Unit after acute intracerebral hemorrhage requiring surgical treatment, mechanical thrombectomy for acute ischemic stroke, embolization of aneurysm causing subarachnoid hemorrhage and scheduled neurosurgical and neuroradiology procedures.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of clevidipine | 1 to 6 hour of clevidipine infusion beginning
  Percentage of patients achieving target systolic blood pressure (SBP)

SECONDARY OUTCOMES:
Incidence of adverse events related to clevidipine treatment | 1 hour after beginning to 24 hours after clevidipine infusion stop
  Tachycardia, atrial fibrillation, hypotension, fever, acute kidney failure, nausea, headache and facial redness.

OTHER OUTCOMES:
Effectiveness of clevidipine treatment according sex | 1 to 6 hours after clevidipine infusion beginning
  Percentage of male and female patients with effective treatment
Effectivennes of clevidipine treatment according medical history | 1 to 6 hours after clevidipine infusion beginning
  Percentage of patients with history of chronic hypertension, ischemic heart disease, stroke, diabetes, hypercholesterolemia, smoking and another cardiovascular risk factor with effective treatment
Effectivennes of clevidipine treatment according neurosurgical procedure | 1 to 6 hours after clevidipine infusion beginning
  Percentage of patients with mechanical thrombectomy, urgent craniotomy, scheduled craniotomy, urgent embolization of aneurysm causing subarachnoidal hemorrhage, urgent embolization of arterio-venous malformations, scheduled embolization of brain aneurysm, intracranial pressure monitoring sensor insertion, intraventricular fibrinolysis, deep brain stimulation for Parkinson's disease with effective treatment
Effectivennes of clevidipine according neurocritical disease | 1 to 6 hours after clevidipine infusion beginning
  Percentage of patients with intracerebral hemorrhage, spontaneous aneurysmal subarachnoid hemorrhage, ischemic stroke, hypertension crisis after scheduled neurosurgery and intracranial hypertension with effective treatment
Effectivennes of clevidipine treatment according poor prognosis factors | 1 to 6 hours after clevidipine infusion beginning
  Percentage of patients with brain hematoma volumes higher than 30 ml, National Institutes Of Health Stroke Scale (NIHSS) higher than 10 points, Fisher scale of aneurysmal subarachnoid hemorrhage of 3 or 4 points and Glasgow Coma Scale less than 8 points with effective treatment
Effectivennes of clevidipine according functional situation | 90 days
  Percentage of patients with modified Rankin scale between 0 to 2 points, 3 to 4 points and 5 to 6 points with effective treatment
Incidence of adverse events according early beginning, first line and effective treatment with clevidipine | 1 hour after beginning to 24 hours after clevidipine infusion stop
  Percentage of patients with early begin of treatment within 24 hours of admission, first line treatment choice, maintenance of goal Systolic Blood Pressure 24 hours after infusion stop and effective treatment presenting any adverse event atributed to clevididipine treatment
Mortality according early beginning, first line and effective treatment with clevidipine | 1 to 90 days
  Percentage of patients with early beginning of clevidipine treatment within 24 hours of admission, first line treatment, maintenance of Systolic Blood Pressure higher than 48 hours and effective treatment dead
Major complications according early beginning, first line and effective treatment with clevidipine | 1 to 15 days
  Percentage of patients with early beginning of clevidipine treatment within 24 hours of admission, first line treatment, maintenance of Systolic Blood Pressure higher than 48 hours and effective treatment presenting major neurological complications like rebleeding, hematoma expansion, brain swelling, intracranial hypertension, vasospasm and neurological deterioration not explained for the above
Hematoma expansion in subgroups | 1 to 7 days
  Percentage of patients with brain hematoma expansion presenting Systolic Blood Pressure higher than 180 mmHg, age higher than 65 years old, Glasgow Coma Scale up to 8 points at admission, chronic hypertension history, intracranial hypertension, subararchnoidal hemorrhage, intraventricular hemorrhage, hematoma volumes higher than 30 ml, spot sign, begin of treatment in first 5 hours of admission, effective treatment and clevidipine as first line.
Vasospasm in subgroups | 1 to 15 days
  Percentage of patients with spontaneous aneurysmal subararachnoid hemorrhage presenting vasospasm with a Systolic Blood Pressure higher than 160 mmHg, Fisher score of 3 to 4 points at admission, effective treatment and clevidipine as first line treatment.
Aneurysm rebleeding in subgroups | 1 to 7 days
  Percentage of patients with rebleeding after spontaneous aneurysmal subarachnoidal hemorrhage presenting Systolic Blood Pressure higher than 160 mmHg, aneurysms of posterior brain circulation, intracranial hypertension, effective treatment and first line treatment with clevidipine

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Escontrela, Consultant, Principal Investigator — Biobizkaia Health Research Institute
Locations (1):
- Biocruces, Barakaldo, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Database